CLINICAL TRIAL: NCT02752048
Title: A Randomized Phase IIa Study of TAS-205 in Patients With Duchenne Muscular Dystrophy
Brief Title: A Phase IIa Study of TAS-205 for Duchenne Muscular Dystrophy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Taiho Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Taiho10053040
Record Dates: First submitted 2016-04-06; First posted 2016-04-26 (Estimated); Results first posted 2020-04-20 (Actual); Last update posted 2020-04-20 (Actual); Status verified 2020-03

CONDITIONS: Duchenne Muscular Dystrophy
MeSH Terms: conditions — Muscular Dystrophy, Duchenne | interventions — TAS-205

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- TAS-205（Low dose group） (Experimental): Low dose group：Oral administration of tablets for 24 weeks, bis in die (BID) after meal The number of tablets of the study drug corresponding to the dosage (6.67-13.33 mg/kg/dose) by body weight within 14 days before enrollment was to be administered within 30 minutes after breakfast and dinner.
  Interventions: Drug: TAS-205
- TAS-205（High dose group） (Experimental): High dose group: Oral administration of tablets for 24 weeks, bis in die (BID) after meal The number of tablets of the study drug corresponding to the dosage (13.33-26.67 mg/kg/dose) by body weight within 14 days before enrollment was to be administered within 30 minutes after breakfast and dinner.
  Interventions: Drug: TAS-205
- Placebo (Placebo Comparator): Placebo group: Oral administration of tablets for 24 weeks, BID after meal
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TAS-205 — 2 groups: Low dose group, High dose group. Oral administration for 24 weeks, bis in die (BID) after meal
  Arms: TAS-205（High dose group）; TAS-205（Low dose group）
Drug: Placebo — 1 group: Placebo group. Oral administration for 24 weeks, BID after meal
  Arms: Placebo

SUMMARY:
The objective of this study is to evaluate the efficacy after 24-week repeated oral doses of TAS-205 in patients with Duchenne Muscular Dystrophy (DMD) in an exploratory manner.

DETAILED DESCRIPTION:
Duchenne Muscular Dystrophy (DMD) is the most common fatal genetic disorder diagnosed in childhood, affecting approximately 1 in 3,500 lives male births. DMD patients suffer from a relentless decline in muscle strength that impairs the ability of walking and breathing, resulting in their lives with wheelchairs and then loss of upper body function. The main objective of this study is to evaluate the efficacy after 24-week repeated oral doses of TAS-205 in patients with DMD in an exploratory manner. The objective of this study is also to evaluate the safety, the dose-response and the urinary excretion of pharmacodynamic (PD) marker after 24-week repeated oral doses of TAS-205 in DMD patients.

ELIGIBILITY:
Inclusion Criteria:

* Able to give an informed consent. If applicable, able to give an informed assent.
* Phenotypic evidence of DMD.
* Male and ≧5 years of age.
* Bodyweight ≧7.5 kg and <60 kg.
* Able to complete the 6MWD test with a distance of at least 75 m.
* Able to take tablets.
* If taking oral glucocorticoids no significant change in the total daily or dosing 6 months before enrollment.

Exclusion Criteria:

* Any serious drug allergy.
* A forced vital capacity (FVC) of <50% of predicted value.
* Wearing a respirator continuously (except for the use during sleep).
* A left ventricular ejection fraction (EF) of <40% or fractional shortening (FS) of <25% on echocardiogram.
* Clinically significant cardiac failure and respiratory failure.
* Ongoing immunosuppressive therapy (other than corticosteroids) .
* Surgical history or plan for surgery that may affect muscular strength or motor function.
* Any injury that may affect muscular strength or motor function.
* With any systemic allergic disease or any chronic inflammatory disease.
* Previous gene therapy (exon skipping, or stop codon read through therapy), cell-based therapy, or any other investigational agents.

Min Age: 5 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2016-05; Primary Completion 2017-05-15 (Actual); Study Completion 2017-10-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Taiho Pharmaceutical Co., Ltd., Study Director — Taiho Pharmaceutical Co., Ltd.
Locations (11):
- Japan (11):
  - Nagoya City University Hospital, Aichi
  - National Hospital Organization Nagara Medical Center, Gifu
  - Kobe University Hospital, Hyōgo
  - National Hospital Organization Utano Hospital, Kyoto
  - Shinshu University Hospital, Nagano
  - National Hospital Organization Niigata National Hospital, Niigata
  - National Hospital Organization Toneyama National Hospital, Osaka
  - National Hospital Organization Higashisaitama Hospital, Saitama
  - Tokyo Women's Medical University Hospital, Tokyo
  - National Center of Neurology and Psychiatry, Tokyo
  - Tottori University Hospital, Tottori

REFERENCES:
- [Derived] Komaki H, Maegaki Y, Matsumura T, Shiraishi K, Awano H, Nakamura A, Kinoshita S, Ogata K, Ishigaki K, Saitoh S, Funato M, Kuru S, Nakayama T, Iwata Y, Yajima H, Takeda S. Early phase 2 trial of TAS-205 in patients with Duchenne muscular dystrophy. Ann Clin Transl Neurol. 2020 Feb;7(2):181-190. doi: 10.1002/acn3.50978. Epub 2020 Jan 20. PMID 31957953

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | TAS-205（Low Dose Group） | TAS-205（High Dose Group） | Placebo
Started | 11 | 12 | 13
Completed | 11 | 12 | 10
Not Completed | 0 | 0 | 3
Not completed — Withdrawal by Subject | 0 | 0 | 3

BASELINE CHARACTERISTICS:
Population: Analysis population was per protocol set. One patients excluded from TAS-205 High dose group, and three excluded from placebo group.
Groups:
- Total: Total of all reporting groups
Arm/Group | TAS-205（Low Dose Group） | TAS-205（High Dose Group） | Placebo | Total
Number analyzed (Participants) | 11 | 11 | 10 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 11 | 11 | 10 | 32
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 11 | 11 | 10 | 32
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 11 | 11 | 10 | 32
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Japan | 11 | 11 | 10 | 32

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline to 24 Weeks in the 6-minute Walk Distance (6MWD)
Description: The distance the subject can walk as fast as possible in 6 minutes will be evaluated.
Time Frame: baseline, 24 weeks
Measure: Mean (Standard Deviation); unit: meter
Arm/Group | TAS-205（Low Dose Group） | TAS-205（High Dose Group） | Placebo
Number analyzed (Participants) | 11 | 11 | 10
meter | -3.5 (67.3) | -7.5 (37.3) | -17.0 (55.6)

2. Secondary Outcome: Mean Change From Baseline in Time to Rise From the Floor
Description: The time required for the subject to rise from a supine position on the floor as quickly as possible will be evaluated.
Time Frame: baseline, and 24 weeks
Measure: Mean (Standard Deviation); unit: second
Arm/Group | TAS-205（Low Dose Group） | TAS-205（High Dose Group） | Placebo
Number analyzed (Participants) | 11 | 11 | 10
second | 4.011 (6.209) | 1.283 (2.547) | 2.633 (4.246)
Statistical Analysis 1: Comparison: TAS-205（Low Dose Group） vs Placebo; Test type: Other — Change in time to rise from the floor from baseline to Week 24 were calculated to evaluate; p = 0.596, t-test, 2 sided; Mean Difference (Final Values) = -1.378, 95% CI 2-sided [-6.757 to 4.000]
Statistical Analysis 2: Comparison: TAS-205（High Dose Group） vs Placebo; Test type: Other — Change in time to rise from the floor from baseline to Week 24 were calculated to evaluate; p = 0.433, t-test, 2 sided; Mean Difference (Final Values) = 1.349, 95% CI 2-sided [-2.220 to 4.918]

3. Secondary Outcome: Mean Change From Baseline in Time to Walk/Run for 10meters
Description: The time required for the subject to run or walk as quickly as possible a 10 m-wide passage with marks affixed on the floor will be evaluated.
Time Frame: baseline, and 24 weeks
Measure: Mean (Standard Deviation); unit: second
Arm/Group | TAS-205（Low Dose Group） | TAS-205（High Dose Group） | Placebo
Number analyzed (Participants) | 11 | 11 | 10
second | 1.113 (1.140) | 1.025 (1.296) | 0.629 (1.272)
Statistical Analysis 1: Comparison: TAS-205（Low Dose Group） vs Placebo; Test type: Other — Change in 10-m walk/run test from baseline to Week 24 were calculated to evaluate; p = 0.382, t-test, 2 sided; Mean Difference (Final Values) = -0.484, 95% CI 2-sided [-1.618 to 0.650]
Statistical Analysis 2: Comparison: TAS-205（High Dose Group） vs Placebo; Test type: Other — Change in 10-m walk/run test from baseline to Week 24 were calculated to evaluate; p = 0.501, t-test, 2 sided; Mean Difference (Final Values) = -0.397, 95% CI 2-sided [-1.610 to 0.817]

4. Secondary Outcome: Mean Change From Baseline in Time to up and go (TUG)
Description: This test will assess the extent of the subject's composite mobility, including standing up, walking, repositioning the body, and balancing.
Time Frame: baseline, and 24 weeks
Measure: Mean (Standard Deviation); unit: second
Arm/Group | TAS-205（Low Dose Group） | TAS-205（High Dose Group） | Placebo
Number analyzed (Participants) | 11 | 11 | 10
second | 0.594 (2.156) | 0.286 (1.626) | 0.061 (1.626)
Statistical Analysis 1: Comparison: TAS-205（Low Dose Group） vs Placebo; Test type: Other — Change in time to up and go from baseline to Week 24 were calculated to evaluate; p = 0.549, t-test, 2 sided; Mean Difference (Final Values) = -0.533, 95% CI 2-sided [-2.363 to 1.298]
Statistical Analysis 2: Comparison: TAS-205（High Dose Group） vs Placebo; Test type: Other — Change in time to up and go from baseline to Week 24 were calculated to evaluate; p = 0.767, t-test, 2 sided; Mean Difference (Final Values) = -0.225, 95% CI 2-sided [-1.801 to 1.351]

ADVERSE EVENTS:
Time Frame: From registration point to the end of follow-up period which was after four weeks from the end of 24-weeks administration
Arm/Group | TAS-205（Low Dose Group） | TAS-205（High Dose Group） | Placebo
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 9/11 | 9/12 | 10/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TAS-205（Low Dose Group） (N=11) | TAS-205（High Dose Group） (N=12) | Placebo (N=12)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Dental caries (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Stomatitis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Peripheral swelling (General disorders) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1) | 2 (2)
Gastroenteritis (Infections and infestations) | 2 (2) | 3 (3) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Impetigo (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Mumps (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia mycoplasmal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 2 (2) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Beta haemolytic streptococcal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Chillblains (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2)
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Blood corticotrophin decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Cortisol decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Glucose urine present (Investigations) | 0 (0) | 1 (1) | 0 (0)
Muscle enzyme increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Cystatin C increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Urobilinogen urine increased (Investigations) | 0 (0) | 2 (2) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 2 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 2 (2)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Head banging (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting psychogenic (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3) | 0 (0)
Dyshidrotic eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Leukoderma (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Palmar erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Papule (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2016-04-07): https://cdn.clinicaltrials.gov/large-docs/48/NCT02752048/Prot_000.pdf
  • Statistical Analysis Plan (2018-08-14): https://cdn.clinicaltrials.gov/large-docs/48/NCT02752048/SAP_001.pdf